CLINICAL TRIAL: NCT06203522
Title: Factors Associated With Successful Completion of MRI in Children Undergoing a Vigil Sedation With Dexmedetomidin: an Observational Study
Brief Title: Factors Associated With Successful Completion of MRI in Children Undergoing a Vigil Sedation With Dexmedetomidin
Acronym: RIDEX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-12'Obs-CHRMT
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Procedural Sedation; EEG; MRI
Keywords: Dexmedetomidin; procedural sedation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI with Dexmedetomidin: Mean age is compared between the "pass" and "fail" groups using a Student's t-test accounting for inequality of variances. MRI success rates are compared between subgroups using Fischer's exact tests. Finally, factors related to MRI success rates are investigated using multivariate logistic regression, including all the factors described above.
  Interventions: Procedure: Data collection of successful completion of MRI

INTERVENTIONS:
Procedure: Data collection of successful completion of MRI — age, sex, autistic disorders, epilepsy, polyhandicap, non-autistic neurodevelopmental disorders, success of MRI procedure

SUMMARY:
This is a retrospective cohort study aiming to determine whether the use of Dexmedetomidine (DEX) to sedate children prior to MRI scanning is more or less effective in children with autism spectrum disorders or other neurodevelopmental disorders compared to other children.

DETAILED DESCRIPTION:
Performing brain MRI on children under 5, or in cases of autism or disability, is often complex. In fact, this examination requires total immobilization of the child for at least 20 minutes. The noise and the fact that the child is lying in a sort of tunnel add to the child's stress.

General anesthesia with propofol is widely used in France, but requires invasive orotracheal intubation or mask ventilation. There are no national or international recommendations for pediatric MRI sedation procedures.

Intranasal dexmedetomidine (DEX) is used for brain MRI, cardiac ultrasound, ophthalmology, dental treatment and brain computed tomography (CT) in patients aged 3 months to 12 years. Its superior efficacy has been demonstrated in a number of studies compared with the most commonly used medicated procedural sedation techniques, but only one study in France has prospectively analyzed the efficacy of DEX IN for performing cerebral MRIs, but without assessing efficacy and tolerance in subgroups of children: with or without neurodevelopmental disorders, epilepsy, autism, age.

ELIGIBILITY:
Inclusion Criteria:

* patients under 18 years of age sedated with DEX IN prior to MRI.

Exclusion Criteria:

* incomplete or missing medical records

Ages: 3 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients under 18 years of age sedated with DEX IN prior to MRI.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Successful Completion of MRI, defined as the radiologist having no reservations about the interpretation of the images. | Immediately after procedure
  Successful Completion of MRI, defined as the radiologist having no reservations about the interpretation of the images (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Charlotte CULLIER, MD, Principal Investigator — CHR Metz Thionville Hopital Mercy
Locations (1):
- CHR Metz-Thionville/Hopital Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No
According to the French law and the French Data Protection Authority (CNIL), it is not possible to share publicly individual participant data, but only their conclusions through peer-reviewed publications and conferences.